CLINICAL TRIAL: NCT06518447
Title: Randomized Cross-clinical Trial Comparing Precision of Conventional Stabilization Splints (Michigan Type) Versus CAD/CAM Splints With Fully Digital Flow
Brief Title: Conventional vs Digital CAD/CAM Splints for Bruxism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 59319422.3.0000.5336
Record Dates: First submitted 2024-07-03; First posted 2024-07-24 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2024-07

CONDITIONS: Bruxism
Keywords: occlusal splints; computer-aided design; bruxism
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant Masking:
  Patients will not be informed whether they are receiving the conventional stabilization splint or the CAD/CAM splint. The splints will be marked with small, inconspicuous letters (A for Group A and B for Group B) during the fabrication process to minimize the possibility of the patients identifying which type of splint they are using. Additionally, both splints will be polished similarly to ensure no noticeable differences in appearance or texture.
  Researcher Masking:
  The primary researcher conducting patient evaluations and data analysis will be blinded to the group assignments. This researcher will not be involved in the fabrication or fitting of the splints, thereby maintaining an objective perspective during assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital occlusal splints (CAD/CAM) (Experimental): Patients in this arm will receive a CAD/CAM occlusal stabilization splint created using a fully digital workflow. The process includes:
  1. Digital Impression: digital scan of the mouth will be performed using a 3shape® intraoral scanner.
  2. Digital Design: The scanned data will be processed using Dental Wings' DWOS® software to design the occlusal splint virtually. The design will ensure the splint follows the Michigan splint type specifications.
  3. Manufacturing: The designed splint will be fabricated using a Straumann® P series rapidshape P30+ 3D printer with a specific acrylic resin, Cosmos Splint. The splint will be polished to ensure comfort and fit, while maintaining the same surface texture as the conventional splint.
  4. Fitting and Adjustment: The digitally fabricated splint will be fitted and adjusted as necessary to ensure proper adaptation and occlusal contacts. An Occlusense device will be used to verify and adjust the occlusal contacts during the fitting process.
  Interventions: Device: Digital occlusal splints (CAD/CAM)
- Conventional occlusal splints (Active Comparator): Patients in this arm will receive a conventional occlusal stabilization splint fabricated using traditional analog methods. The process includes:
  1. Impression Taking: Impressions of the patient's upper and lower arches will be taken using alginate.
  2. Model Preparation: The plaster models will be mounted on a semi-adjustable articulator using a centric relation occlusal record. A wax-up of the occlusal splint will be created following the Michigan splint type specifications.
  3. Manufacturing: The wax-up will be processed and flasked with heat-cured acrylic resin to create the final splint. The splint will be polished similarly to the digital splint to ensure a consistent appearance and texture.
  4. Fitting and Adjustment: The conventional splint will be fitted and adjusted to ensure proper adaptation and occlusal contacts. An Occlusense device will be used to verify and adjust the occlusal contacts during the fitting process.
  Interventions: Device: Conventional occlusal splints

INTERVENTIONS:
Device: Digital occlusal splints (CAD/CAM) — Consists of occlusal stabilization intra-oral splints fabricated using a fully digital workflow, involving intraoral scanning, virtual design, and 3D printing to ensure precise fit and comfort.
  Other Names: Digital intra-oral device
  Arms: Digital occlusal splints (CAD/CAM)
Device: Conventional occlusal splints — Consists of occlusal stabilization splints fabricated using traditional analog methods, including physical impressions, plaster models, and manual processing with heat-cured acrylic resin to achieve the desired occlusal arrangement.
  Other Names: Conventional intra-oral device
  Arms: Conventional occlusal splints

SUMMARY:
This is a randomized controlled trial with a crossover design, which intends to enroll 20 adult patients aged between 20 and 55 years with confirmed or probable sleep bruxism. Participants will be randomized to receive either a conventional stabilization splint or a CAD/CAM splint. Each patient will use one type of splint for 30 days, followed by a 15-day wash-out period, after which they will switch to the other type of splint. The study aims to compare the quality, precision, and comfort of the two types of occlusal splints. Outcomes will include manufacturing time, amount of in-mouth adjustments, adaptation, occlusal contacts, and participant satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged between 20 and 55 years.
* Probable or confirmed diagnosis of sleep bruxism.
* No previous treatment with occlusal splints.
* Absence of periodontal diseases and/or dental fractures.
* Patients must have a minimum of 28 teeth.

Exclusion Criteria:

* Patients with systemic diseases affecting the temporomandibular joint, such as rheumatoid arthritis, osteoarthritis, and osteoporosis.
* Chronic users of medications that may interfere with the study results, including analgesics, anti-inflammatory drugs, anxiolytics, antidepressants, and anticonvulsants.
* Patients with a history of temporomandibular joint surgery.
* Pregnant or breastfeeding women.
* Patients with severe dental misalignment or malocclusion that would affect splint fitting and evaluation.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of occlusal contacts | Immediately after the initial installation
  The number of occlusal contacts will be measured using the OccluSense® device

SECONDARY OUTCOMES:
Time Required for Splint Adjustment | Immediately after the initial installation and adjustment
  The time required to adjust each splint during the fitting process
Participant satisfaction after installation | Immediately after the initial installation and adjustment
  Patients will assess their overall satisfaction with the splints using a 5-point Likert scale, with 1 meaning the lowest score of satisfaction and 5 meaning the highest score of satisfaction.
Participant satisfaction after 30 days | After 30 days of use
  Patients will assess their overall satisfaction with the splints using a 5-point Likert scale, with 1 meaning the lowest score of satisfaction and 5 meaning the highest score of satisfaction.
Splint comfort after installation | Immediately after the initial installation and adjustment
  Patients will assess comfort with the splints using a 5-point Likert scale, with 1 indicating the lowest level of comfort and 5 indicating the highest level of comfort.
Splint comfort after 30 days | After 30 days of use
  Patients will assess comfort with the splints using a 5-point Likert scale, with 1 indicating the lowest level of comfort and 5 indicating the highest level of comfort.
Splint stability after installation | Immediately after the initial installation and adjustment
  Patients will assess the stability of the splints (retention) during use using a 5-point Likert scale, with 1 indicating the lowest level of stability (frequent movement) and 5 indicating the highest level of stability (no movement).
Splint stability after 30 days | After 30 days of use
  Patients will assess the stability of the splints (retention) during use using a 5-point Likert scale, with 1 indicating the lowest level of stability (frequent movement) and 5 indicating the highest level of stability (no movement).

CONTACTS AND LOCATIONS:
Overall Officials: Marcio L Grossi, PhD, Study Chair — Pontifícia Universidade Católica do Rio Grande do Sul
Locations (1):
- Faculdade de Odontologia. Pontifícia Universidade Católica do Rio Grande do Sul., Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No
Not planned. Sharing of anonymized data may be considered under exceptional circumstances through direct contact with investigators.